CLINICAL TRIAL: NCT07166250
Title: Comparison of the Effects of Quadratus Lumborum Block and Retrolaminar Block on Postoperative Pain in Lumbar Disc Herniation Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nermin Kandemir, research assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KANDEMIR-QLB-O
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Herniation; Postoperative Pain
Keywords: Quadratus Lumborum Block; Retrolaminar Block; Spine Surgery Analgesia; Opioid Consumption
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial comparing quadratus lumborum block and retrolaminar block in patients undergoing lumbar disc herniation surgery.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Experimental): Patients randomized to this group will receive an ultrasound-guided quadratus lumborum block (QLB) with local anesthetic injection before surgical incision for postoperative pain management.
  Interventions: Procedure: Quadratus Lumborum Block
- Retrolaminar Block (Experimental): Patients randomized to this group will receive an ultrasound-guided retrolaminar block (RLB) with local anesthetic injection before surgical incision for postoperative pain management.
  Interventions: Procedure: Retrolaminar Block

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Ultrasound-guided quadratus lumborum block performed preoperatively using local anesthetic injection at the thoracolumbar fascia for postoperative analgesia in lumbar disc herniation surgery.
  Arms: Quadratus Lumborum Block
Procedure: Retrolaminar Block — Ultrasound-guided retrolaminar block performed preoperatively using local anesthetic injection into the retrolaminar space for postoperative analgesia in lumbar disc herniation surgery
  Arms: Retrolaminar Block

SUMMARY:
This study aims to compare the analgesic efficacy of quadratus lumborum block (QLB) and retrolaminar block (RLB) in patients undergoing lumbar disc herniation surgery. Both regional anesthesia techniques are increasingly used for postoperative pain management, but there is limited evidence directly comparing their effectiveness. The primary outcome is the postoperative pain score, while secondary outcomes include opioid consumption and patient satisfaction.

DETAILED DESCRIPTION:
Effective postoperative pain management is essential in patients undergoing lumbar disc herniation surgery. Regional anesthesia techniques, such as quadratus lumborum block (QLB) and retrolaminar block (RLB), have been increasingly used as alternatives or adjuncts to systemic analgesics. QLB provides analgesia by targeting the thoracolumbar fascia and spreading to the paravertebral space, whereas RLB is considered a simpler and potentially safer approach with similar analgesic potential.

This randomized controlled clinical trial is designed to compare the efficacy and safety of QLB and RLB for postoperative pain control. Adult patients scheduled for elective lumbar disc herniation surgery under general anesthesia will be randomized into two groups. One group will receive ultrasound-guided QLB, and the other group will receive ultrasound-guided RLB before surgical incision.

The primary outcome is postoperative pain intensity measured using a numerical rating scale (NRS) at multiple time intervals within the first 24 hours after surgery. Secondary outcomes include total opioid consumption, time to first analgesic request, incidence of block-related complications, and overall patient satisfaction. The results of this study are expected to provide evidence for the optimal regional technique for postoperative analgesia in lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-65 years American Society of Anesthesiologists (ASA) physical status I-II-III Scheduled for elective lumbar disc herniation surgery under general anesthesia Willing to participate and provide written informed consent Patients scheduled for elective lumbar disc herniation surgery

Exclusion Criteria:

Patients requiring emergency surgery ASA physical status classification IV-V Known coagulopathy Ongoing anticoagulant therapy History of allergy to local anesthetics Localized infection at the block injection site Presence of spinal, paraspinal, or regional deformities at the block area Inability to understand or use the verbal pain rating scale Chronic use of analgesic medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity (NRS score) | Within the first 24 hours after surgery
  Pain intensity will be assessed using the Numerical Rating Scale (0-10) at rest and during movement.

SECONDARY OUTCOMES:
Total opioid consumption | 24 hours after surgery
  Total amount of opioid analgesics (morphine equivalent) administered in the first 24 hours postoperatively.
Time to first analgesic request | 24 hours after surgery
  Time interval between the end of surgery and the first request for additional analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: dilek icli, prof. dr., Principal Investigator — Kocaeli University, Department of Anesthesiology and Reanimation
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No